CLINICAL TRIAL: NCT07332260
Title: Alzheimer's Disease and Faecal Microbiota Transplantation
Brief Title: Alzheimer's Disease and Faecal Microbiota Transplantation -a Pilot Study
Acronym: AD-FMT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 853867/2025
Record Dates: First submitted 2025-11-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer s Disease; Faecal Microbiota Transplantation (FMT)
Keywords: Alzheimer's disease; Dementia; Gut microbiota; faecal microbiota transplantation; FMT
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Single-arm, single-centre, non-randomised, open label intervention study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Faecal microbiota transplantation (FMT) (Experimental): Single-group, single-centre, open-label. Intervention: Faecal microbiota transplantation administered via colonoscopy to the right side of the colon.
  Interventions: Biological: Biological: Preprocessed thawed donor FMT

INTERVENTIONS:
Biological: Biological: Preprocessed thawed donor FMT — Biological: Preprocessed FMT solution is administered to the right side of the colon during a colonoscopy.

SUMMARY:
The goal of this study is to assess the feasibility and safety of faecal microbiota transplantation for Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia.

Studies suggest that the gut flora may play a role in the development and/or progression of AD. The gut flora is found to be different in AD compared to healthy individuals. There is also support for a link between the gut flora and diseases affecting the brain, including AD.

Stool transplantation is an established medical treatment for Clostridioides difficile infections by restoring the balance of the gut flora. In this study, gut flora (a stool solution) is transferred from a healthy individual to an individual with AD. The stool transplantation is given during a colonoscopy examination of the large bowel.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's dementia mild to moderate stage
* Presence of Alzheimer pathology core 1 biomarkers as defined by National Institute on Aging-Alzheimer's Association (NIA-AA) criteria (2024)
* Capable of giving informed consent

Exclusion Criteria:

* Contraindications for colonoscopy examination
* Contraindications for Magnetic Resonance Imaging (MRI)
* Life expectancy < 1 year
* Clinical frailty scale 7 or more
* History of seizure disorder
* History of brain tumour or intracranial bleed
* Major psychiatric disorder such as schizophrenia, bipolar disorder, or major depressive disorder
* Alcohol or substance abuse
* Decompensated heart disease
* Malignancy
* Current use of anticoagulant treatment (dual acting oral anticoagulant or warfarin)
* Pregnant or planning pregnancy
* Colonic adenomas over 1 cm, tumours or signs of active colitis on colonoscopy
* Status after colectomy or hemicolectomy
* Inflammatory bowel disease
* Immunocompromised individual
* Receiving biological/antibody treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events and serious adverse events. [Safety] | From baseline to 3 months after faecal microbiota transplantation
  Incidence of adverse events (AE) and serious adverse events (SAE). AE and SAE are evaluated by review of the medical record, questions of AE and SAE in person or by telephone, and AE and SAE forms.
Rate of participant recruitment [Feasibility] | 1 year
  Number of weeks needed to include ten participants for study intervention group
Number participants that complete colonoscopy [Feasibility] | 1 year
  Number of participants that complete colonoscopy
Time used per intervention [Feasibility] | 1 year
  Time given in hours and minutes of total time used for intervention per participant including colonoscopy and faecal microbiota transplantation.
Number that meet study eligibility [Feasibility] | 1 year
  Number of participants who are screened for study eligibility. Number who meet inclusion and exclusion criteria.
Number that complete study [Feasibility] | Baseline and 3 months after study intervention
  Proportion of participants enrolled that complete the study follow-up.
Engraftment of faecal microbiota transplantation (FMT) | baseline and 3 months after study intervention
  Comparison of the taxonomic composition of the microbiome in participants faecal samples at baseline and 3 months after FMT, with donor faecal sample. Metagenomic sequencing of faecal samples will be used.

SECONDARY OUTCOMES:
Cognition: Clinical dementia rating scale - sum of boxes (CDR-SB) | Baseline and 3 months after study intervention
  Clinical Dementia Rating Scale- Sum of Boxes (CDR-SB) is a cognitive test that is used to assess the severity of dementia. It evaluates six cognitive and functional domains, where the scores are summed to provide a total score from 0 to 18. It is useful for tracking disease progression.
  Participants will be tested at baseline and 3 months after faecal microbiota transplantation.
Cognition: Montreal Cognitive Assessment (MoCA) | Baseline and 3 months after study intervention
  Change in the Montreal Cognitive Assessment (MoCA) from baseline and 3 months after intervention. The MoCA is a brief cognitive test used to detect mild cognitive impairment and early stages of dementia. It is scored out of 30 points. A lower score indicates a higher impairment.
Cognition: Trailmaking Test (TMT | Baseline and 3 months after study intervention
  Change in Trailmaking Tests (TMT) comparing baseline and 3 month after study intervention. The TMT is a neuropsychological test in two parts where visual attention, visuomotor coordination, processing speed and executive function are tested. The test is performed in two parts (A and B) and the result is reported in seconds used to complete task.
Cognition: Wordlist | Baseline and 3 months after study intervention
  Change in verbal memory assessed by the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) comparing baseline and 3 months after study intervention. The CERAD wordlist is a standard test where the participant is asked to recall a list of ten words. Its result is given as number of words correctly recalled, adjusted to normative data.
Cognition: neuropsychiatric inventory (NPI) | Baseline and 3 months after study intervention
  Change in neuropsychiatric inventory (NPI) will be assessed comparing baseline with 3 months after study intervention.
  The NPI is a questionnaire following interview with a caregiver or informant who is familiar with the participant. Results are given as a number scale from 0-12 across the behavioural and psychological domains commonly affected in dementia. The domain scores are added up to a total NPI score which can range from 0 to 144. A higher NPI score indicates a greater neuropsychiatric symptom burden.
Cognition: Activities of Daily Living (ADL) | Baseline and 3 months after study intervention
  Changes in activities of daily living (ADL) will be assessed comparing baseline and 3 months after study intervention. ADL will be measured by a number score for instrumental and personal activities of living using standardised questionnaires.
  ADL is given as a score, a lower score indicates impairment.
Changes in Quality of Life | Baseline and 3 months after intervention
  Changes in Quality of Life at baseline and 3 months after study intervention will be assessed using the questionnaire EuroQol-5-Dimensions (EQ-5D) which is a standardised test where an individual rates their health-related quality of life based on five dimensions as well as a scale from 0 (worst imaginable health) to 100 (best imaginable health).

OTHER OUTCOMES:
Changes in biomarkers for Alzheimer's disease | Baseline and 3 months after intervention
  Comparison of plasma phosphorylated tau at threonine 217 (p-tau217) levels measured at baseline and 3 months after study intervention will be compared.
  P-tau217 is a specific biomarker and a core biomarker for Alzheimer's disease. It is measured in picograms per milliliter.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Dixon Gundersen, MBChB, PhD, Principal Investigator — University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: No